CLINICAL TRIAL: NCT06682754
Title: Use of Balance Detection Devices for Elderly People Under the Influence of Stress (DEPIE)
Brief Title: Detection of Balance in the Elderly Under the Influence of Stress
Acronym: DEPIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: European Union (Other); Castilla-La Mancha Health Service (Other)
Responsible Party: Principal Investigator, Susana Nunez Nagy, PhD. Associate Professor., University of Alcala
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CEIP/2023/5/110
Record Dates: First submitted 2024-10-31; First posted 2024-11-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Balance

STUDY DESIGN:
Masking Description: Although all participants will perform the same intervention, they will not know which intervention the other participants are performing. In addition, the entire experimental session (both baseline and experimental test) is computerized, so the researcher in charge of the experiment will only ensure that all systems are working properly. On the other hand, the outcome evaluator will analyze the baseline and experimental moments without knowing whether the data belong to one or the other moment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All participants will perform a baseline and an experimental test. There will be a group of young people and a group of older people, but all participants will perform the same intervention
  Interventions: Other: Stress

INTERVENTIONS:
Other: Stress — All participants will perform a baseline test in which they will first be asked to visualize low-arousal IAPS images for three minutes while seated in a chair, and then get up, walk to a table with two bottles, transfer liquid from one bottle to the other, return to the starting chair and sit down again. Subsequently, they will perform an experimental test, where they will repeat the same movements as in the baseline test after visualizing high-arousal IAPS images for three minutes. In addition, IAPS images will continue to be projected in the background while participants perform the described motor tasks.

SUMMARY:
The aging process involves physiological changes in organs and tissues that can evolve towards fragility and increased risk of falls. Falls, which can be one of the adverse results of frailty in older people, are the second leading cause of death worldwide. When an elderly person falls, it entails not only hospitalization, immobilization, and the consequent deterioration, but also usually causes fear of falling again, which can also lead to the onset of disability. The inherent aging process can be linked to the deterioration of postural control and balance, posing serious health problems. In falls in the elderly, both sensorimotor and cognitive functions are affected, the functioning of which is degraded to a greater extent by anxiety and stress. Nowadays, more extensive, and more precise research is needed in the study of the interactions between cognition, stress, and postural control in the context of postural instability and falls in older adults.

The purpose of the DEPIE Project is to detect whether neuromuscular changes that occur when exposed to stressful situations can affect the postural and motor control of the elderly.

To this end, all participants will undergo the same intervention. Firstly, they will all take a baseline cognitive and physical assessment. Afterwards, they will take the experimental session, which will consist of a baseline test and an experimental test. During the baseline test, participants will visualize International Affective Picture System (IAPS) images of low arousal and during the experimental test of high arousal. Finally, physical assessment tests will be repeated.

Young and older adults will be tested. Additionally, sub-analyses will be conducted within the elderly group differentiating the degree of cognitive impairment and functional dependence.

The primary outcome measures will be surface electromyography, pressures on the floor, activity on manipulation, and balance.

The secondary outcome measures will be heart rate variability, respiratory rate and the visual analogue scale on unease after visualisation of the images.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (ages 18-39).
* Older adults (≥65).
* Voluntarily participate in the study.
* Not meeting the exclusion criteria

Exclusion Criteria:

* Any disease, injury, or previous trauma that contraindicates muscular exertion, balance exercises, and/or walking.
* Any physical or mental illness that contraindicates exposure to stimuli generating emotional stress, such as severe depression or severe psychosis
* Difficulties in understanding study information and providing informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pressures on the floor | It will be assessed while performing the movements of getting up from the chair, walking, manipulating the bottles, returning to the chair and sitting down, both during the baseline test and during the experimental test
  They will be measured by a sensorised blanket that will give information on weight distribution and movement behaviour
Triaxial accelerometry: acceleration and deceleration in object handling | It will be assessed while performing the bottle manipulation movement (during which liquid has to be transferred from one bottle to another), both during the baseline test and during the experimental test
  The maximum acceleration value during the handling activity of two bottles shall be measured with sensors installed on the bottles.
RMS value of the EMG signal | It will be assessed while performing the movements of getting up from the chair, walking, manipulating the bottles, returning to the chair and sitting down, both during the baseline test and during the experimental test
  The root mean square (RMS) value of the EMG signal reflects the level of muscle activation during activity.
EMG: Synchronisation of activation between muscle groups | It will be assessed while performing the movements of getting up from the chair, walking, manipulating the bottles, returning to the chair and sitting down, both during the baseline test and during the experimental test
  It will assess in milliseconds the ability of the muscles to work in a synchronised manner.
EMG: Activation ratio between upper and lower body muscles | It will be assessed while performing the movements of getting up from the chair, walking, manipulating the bottles, returning to the chair and sitting down, both during the baseline test and during the experimental test
  RMS ratio between different muscles
EMG: Median Frequency (MDF) | It will be assessed while performing the movements of getting up from the chair, walking, manipulating the bottles, returning to the chair and sitting down, both during the baseline test and during the experimental test
  In the frequency domain, this median frequency of the EMG signal will be calculated.
Balance | Before the baseline test and after the experimental test
  It will be assessed by Timed Up and Go Test (TUG) and Functional Reach Test (FRT)

SECONDARY OUTCOMES:
Heart Rate Variability | It will be assessed during the visualization of IAPS images both during the baseline test and during the experimental test
  It will be explored for measures of autonomic nervous system activation
Respiratory Rate | It will be assessed during the visualization of IAPS images both during the baseline test and during the experimental test
  It will be explored for measures of autonomic nervous system activation
Analog Visual Scale | Immediately after the baseline test and the experimental test respectively
  It will assess the feeling of unease after performing the baseline test and the experimental test respectively. The scale consists of a line from 0 (= totally relaxed) to 10 (=the most uneasy or restless feeling you have ever felt), which participants have to mark according to their feelings at that moment. Higher scores will correspond to a greater sense of unease.

CONTACTS AND LOCATIONS:
Overall Officials: Susana N Núñez, PhD. Associate Professor, Principal Investigator — University of Alcalá; Bernardo A Alarcos, PhD. Full Professor, Principal Investigator — University of Alcalá
Locations (1):
- University of Alcalá, Alcalá de Henares, Spain

REFERENCES:
- [Derived] Membership of GITES; Alarcos B, Diaz-Pulido B, Fernandez O, Fernandez-Guinea S, Garcia Herraiz A, Lendinez-Chica MDM, Martinez Muela J, Nunez-Nagy S, Perez-Martin Y, Rodriguez-Costa I, Rubio Gonzalez GM, Trapero-Asenjo S, Velasco JR. Detection of balance in the elderly under the influence of stress (DEPIE): A cross-sectional study protocol. PLoS One. 2026 Jan 27;21(1):e0341744. doi: 10.1371/journal.pone.0341744. eCollection 2026. PMID 41592138